CLINICAL TRIAL: NCT06675578
Title: Non Surgical Treatment Using Tulsi Gel Versus Chlorhexidine Gel as Adjunctive in Treatment of Advanced Periodontitis ( Stage III and Stage IV )
Brief Title: Treatment of Periodontitis by Tulsi Gel
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa Gamal Elsayed Mohamed Saleh, Dentist, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-ME-24-12
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Advanced Periodontitis; Stage III Periodontitis; Stage IV Periodontitis
Keywords: periodontitis; clinical attachment loss; advanced periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tulsi Gel group (Active Comparator): Ocimum sanctum
  Interventions: Drug: Tulsi gel
- Chlorhexidine Gel group (Active Comparator): Chlorhexidine
  Interventions: Drug: Chlorhexidine gel

INTERVENTIONS:
Drug: Tulsi gel — After scaling and root debridement, 4% of Tulsi gel will be injected in to the sulcus until it over flooded, at base line, then after one month.
  Other Names: Basil gel
  Arms: Tulsi Gel group
Drug: Chlorhexidine gel — After scaling and root debridement, 1% of Chlorhexidine gel will be injected in to the sulcus until it over flooded, at base line, then after one month.
  Other Names: Corsodyl 1% w/w dental gel
  Arms: Chlorhexidine Gel group

SUMMARY:
This study will be carried out to compare between the effect of 4%Tulsi gel and 1%Chlorohexidine gel as locally administered agents in the treatment of advanced periodontitis. Clinical parameters measurements, microbiological and radiographic assessment will be performed at base line, one month and 3 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in this study will be having advancedI Periodontitis
* Aging from 30 to 50 years old
* Free from any local or systemic risk factors that may affect the results of the study.

Exclusion Criteria:

* Long-term therapy with medications within a month prior to enrollment that could affect periodontal status or healing.
* Pregnant woman and lactating mothers.
* Patients with previous periodontal treatment including scaling and root planning and periodontal surgery in the last 3 and 6 months, respectively.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Clinical parameters | 3 months after end of treatment
  Improvement of the clinical attachment loss in millimeters.
Clinical parameters | 3 months after end of treatment
  Improvement of gingival index.
Clinical parameters | 3 months after end of treatment
  Improvement of probing depth in millimeters.

SECONDARY OUTCOMES:
Microbiological assessment | 3 months after end of treatment
  Counting microbial colony of Porphyromonas gingivalis
Microbiological assessment | 3 months after end of treatment
  Counting microbial colony of Fusobacterium nucleatum
Microbiological assessment | 3 months after end of treatment
  Counting microbial colony of Tannerella forsythia

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al-Azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided